CLINICAL TRIAL: NCT02604823
Title: Efficacy and Safety of Peginterferon Alfa-2a (40 KD) (Pegasys®) in Patients With HBeAg-Positive Chronic Hepatitis B
Brief Title: A Study of Peginterferon Alfa-2a (Pegasys) in Participants With Hepatitis B E-Antigen (HBeAg)-Positive Chronic Hepatitis B Virus (HBV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17700
Record Dates: First submitted 2015-11-04; First posted 2015-11-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

ARMS (3):
- Group A (Naïve Participants) (Experimental): Participants who never received any HBV treatment, will receive peginterferon alfa-2a (180 micrograms [mcg]) subcutaneously once weekly for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a
- Group B (Conventional Interferon Pretreated Participants) (Experimental): Participants who received conventional interferon treatment and had relapse or did not respond, will receive peginterferon alfa-2a (180 mcg) subcutaneously once weekly for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a
- Group C (Lamivudine Pretreated Participants) (Experimental): Participants who received lamivudine and had relapse or did not respond, will receive peginterferon alfa-2a (180 mcg) subcutaneously once weekly for 48 weeks.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a will be administered at a dose of 180 mcg subcutaneously once weekly for 48 weeks.
  Other Names: Pegasys

SUMMARY:
This is a study of the efficacy and safety of peginterferon alfa-2a (Pegasys) in naive, interferon- or lamivudine-pretreated participants with HBeAg-positive chronic HBV. Following 48 weeks treatment, there will be a 24 week period of treatment-free follow-up. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants between 18 to 65 years of age
* HBeAg-positive chronic HBV
* Treatment-naive, or have received and have not responded to or have relapsed on either conventional interferon or lamivudine therapy.

Exclusion Criteria:

* Antiviral or interferon-based therapy for chronic HBV within 6 months of enrollment
* Co-infection with active hepatitis A, C or D virus or with human immunodeficiency virus (HIV)
* Evidence of decompensated liver disease
* Medical condition associated with chronic liver disease other than viral hepatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2003-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with HBV deoxyribonucleic acid (DNA) less than (<) 100,000 copies per milliliters (copies/mL) | 72 weeks
Percentage of participants with HBeAg seroconversion | 72 weeks

SECONDARY OUTCOMES:
Number of participants who achieved HBV DNA levels below limit of detection | Weeks 48 and 72
Number of participants with HBsAg loss | Weeks 48 and 72
Number of participants with both Hepatitis B Surface Antigen (HBsAg) loss and presence of Anti-HBs | Weeks 48 and 72
Number of participants with alanine aminotransferase (ALT) normalization | Weeks 48 and 72
Number of participants with combined response (HBV DNA <100,000 copies/mL, HBeAg loss, and ALT normalization) | Weeks 48 and 72
Incidence of adverse events | up to 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (3):
- China (3):
  - Beijing
  - Guangzhou
  - Shanghai